CLINICAL TRIAL: NCT04802252
Title: A Diagnostic Study of Abnormal Acoustic Waves in Modern Pulse in Benign Prostatic Hyperplasia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Lili Cao, dean of orthopedic department, Qianfoshan Hospital
Other Study IDs: SFUYIN-04
Record Dates: First submitted 2021-03-14; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Benign Prostatic Hyperplasia; Radial Artery
Keywords: Benign prostatic hyperplasia; Sound Waves; Radial Artery; Diagnostic test
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 62 patients with benign prostatic hyperplasia in the experimental group: The pulse sound waves of three parts and five layers of each of the two hands of 62 patients with benign prostatic hyperplasia were collected by acoustic pulse detection system.
- 62 relatively healthy men without benign prostatic hyperplasia in the control group: The pulse sound waves of three parts and five layers of each of the two hands of 62 relatively healthy men without benign prostatic hyperplasia were collected by acoustic pulse detection system.

SUMMARY:
Pulse diagnosis is one of the traditional diagnostic methods of traditional Chinese medicine, which is of great significance in the process of disease diagnosis.Pulse diagnosis is the diagnosis of disease by touching the pulse of the radial artery at the wrist. Different diseases reflect different pulse characteristics.What we've found in long-term clinical observation is that patients with benign prostatic hyperplasia have something different in their pulse,the abnormal pulse we called "astringent pulse".There is no modern physiologic and pathological description on the occurrence of "astringent pulse" in traditional pulse science, so we study it from acoustics perspective.Our team thinks that every beat of the heart produces a vibration, which produces sound waves，the sound waves travel through the blood and eventually reflect off the arterial walls.When an organ(such as the prostate)，develops hyperplasia, local blood flow changes,the flow of blood, which should be laminar, changes and becomes turbulent，the conduction of sound waves in turbulence is disordered，so we end up with pulse features that are different from normal people that are reflected on the arterial wall.

We have previously studied the pulse characteristics of chronic gastritis, coronary heart disease, cirrhosis and some other diseases，different pulse sounds were collected and analyzed using an independently developed Acoustic Pulse Detection System，the ideal results have been obtained.We found that most of the abnormal sound waves were between 20Hz and 500Hz, so we classified this sound wave as low frequency and audible sound wave.Based on the above analysis, this study will use the acoustic pulse detection system to collect the pulse images of patients with benign prostatic hyperplasia(BPH).We expected to collect the pulse waves of 62 patients and 62 relatively healthy people without BPH, and use Fourier transform, wavelet analysis and other analysis methods to study the characteristics of the collected sound waves, and observe the pulse characteristics of BPH disease.Then diagnostic tests were carried out to calculate the sensitivity and specificity of the acoustic pulse detection system in the diagnosis of BPH.

This experiment will further verify the effectiveness of pulse diagnosis of diseases, and finally lay a foundation for the development of pulse diagnostic instrument can diagnose a variety of diseases.

ELIGIBILITY:
Inclusion Criteria:

Test group:

1. From March 2020 to June 2021, patients of Chinese Medicine outpatient department, ward and physical examination were continuously recruited in the First Affiliated Hospital of Shandong First Medical University;
2. Research site: The First Affiliated Hospital of Shandong First Medical University;
3. Comprehensive evaluation of symptoms, signs and ultrasound examination, meeting the diagnostic criteria of BPH in middle-aged and elderly male patients;
4. Ages ranged from 50 to 80 years, and vital signs were stable;
5. Patients with informed consent to accept this pulse collection;

Control group:

1. From March 2020 to June 2021, patients of Chinese Medicine outpatient department, ward and physical examination were continuously recruited in the First Affiliated Hospital of Shandong First Medical University ;
2. Research site: The First Affiliated Hospital of Shandong First Medical University;
3. Symptoms, signs and ultrasonography were evaluated comprehensively, and middle-aged and elderly men with BPH disease were clearly excluded;
4. Ages ranged from 50 to 80 years, and vital signs were stable;
5. Patients with informed consent to accept this pulse collection;

Exclusion Criteria:

Test group:

1. Those who have a serious illness and sit for less than 10 minutes in a quiet state;
2. Symptoms, signs and ultrasonography were evaluated comprehensively, and middle-aged and elderly men with BPH disease were clearly excluded;
3. Patients with severe infectious diseases;
4. Fanguan pulse, oblique flying pulse, etc. who are not easy to collect pulse;
5. Those who have incomplete information due to subjective or objective reasons that affect the result judgment;
6. Patients with Parkinson's or other limb tremors;
7. Those who has not signed an informed consent form;
8. Patients with atrial fibrillation.

Control group:

1. Those who have a serious illness and sit for less than 10 minutes in a quiet state;
2. Comprehensive evaluation of symptoms, signs and ultrasound examination, meeting the diagnostic criteria of BPH in middle-aged and elderly male patients；
3. Patients with severe infectious diseases;
4. Fanguan pulse, oblique flying pulse, etc. who are not easy to collect pulse;
5. Those who have incomplete information due to subjective or objective reasons that affect the result judgment;
6. Patients with Parkinson's or other limb tremors;
7. Those who has not signed an informed consent form;
8. Patients with atrial fibrillation.

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Middle-aged and older men with benign prostatic hyperplasia & middle-aged and older men without benign prostatic hyperplasia
Sampling Method: Non-Probability Sample
Enrollment: 124 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
The characteristic sound waves extracted from radial artery of patients with benign prostatic hyperplasia and relatively healthy men without benign prostatic hyperplasia are distinguished. | 30 minutes
  This characteristic sound wave can distinguish patients with benign prostatic hyperplasia from relatively healthy men without benign prostatic hyperplasia.

CONTACTS AND LOCATIONS:
Overall Officials: Lucheng Song, Doctor, Principal Investigator — The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital
Locations (1):
- Qianfoshan Hospital, The First Hospital affiliated of Shandong First Medical University, Jinan, Shandong, China

REFERENCES:
- [Background] Foo KT. What is a disease? What is the disease clinical benign prostatic hyperplasia (BPH)? World J Urol. 2019 Jul;37(7):1293-1296. doi: 10.1007/s00345-019-02691-0. Epub 2019 Feb 25. PMID 30805683
- [Background] Descazeaud A, Robert G, Delongchamps NB, Cornu JN, Saussine C, Haillot O, Devonec M, Fourmarier M, Ballereau C, Lukacs B, Dumonceau O, Azzouzi AR, Faix A, Desgrandchamps F, de la Taille A; Comite des troubles mictionnels de l'homme de l'association francaise d'urologie. [Initial assessment, follow-up and treatment of lower urinary tract symptoms related to benign prostatic hyperplasia: guidelines of the LUTS committee of the French Urological Association]. Prog Urol. 2012 Dec;22(16):977-88. doi: 10.1016/j.purol.2012.10.001. Epub 2012 Nov 6. French. PMID 23178093
- [Background] Van Asseldonk B, Barkin J, Elterman DS. Medical therapy for benign prostatic hyperplasia: a review. Can J Urol. 2015 Oct;22 Suppl 1:7-17. PMID 26497339
- [Background] Lima CB, Angrimani DSR, Flores RB, Vannucchi CI. Endocrine, prostatic vascular, and proapoptotic changes in dogs with benign prostatic hyperplasia treated medically or surgically. Domest Anim Endocrinol. 2021 Apr;75:106601. doi: 10.1016/j.domaniend.2020.106601. Epub 2020 Nov 23. PMID 33333452
- [Background] Egan KB. The Epidemiology of Benign Prostatic Hyperplasia Associated with Lower Urinary Tract Symptoms: Prevalence and Incident Rates. Urol Clin North Am. 2016 Aug;43(3):289-97. doi: 10.1016/j.ucl.2016.04.001. PMID 27476122
- [Background] Thaler L, Goodale MA. Echolocation in humans: an overview. Wiley Interdiscip Rev Cogn Sci. 2016 Nov;7(6):382-393. doi: 10.1002/wcs.1408. Epub 2016 Aug 19. PMID 27538733
- [Background] Bilton K, Hammer L, Zaslawski C. Contemporary Chinese pulse diagnosis: a modern interpretation of an ancient and traditional method. J Acupunct Meridian Stud. 2013 Oct;6(5):227-33. doi: 10.1016/j.jams.2013.04.002. Epub 2013 Apr 24. PMID 24139459
- [Background] Wang D, Zhang D, Lu G. An Optimal Pulse System Design by Multichannel Sensors Fusion. IEEE J Biomed Health Inform. 2016 Mar;20(2):450-9. doi: 10.1109/JBHI.2015.2392132. Epub 2015 Jan 15. PMID 25608317